CLINICAL TRIAL: NCT06442501
Title: Pregnancy Monkeypox Cohort Study in the South Kivu Province in the DRC
Brief Title: Observational Mondkeypox Pregnancy Cohort
Acronym: PREGMPOXCO
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Colebunders (Other)
Collaborators: Patrick Kototo (Unknown)
Responsible Party: Sponsor-Investigator, Robert Colebunders, Prof, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Other Study IDs: University of Antwerp
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Monkey Pox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin and mucosal swabs, blood, placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPXV infected pregnant women: MPXV infected pregnant women
  Interventions: Other: routine care
- Not MPXV infected pregnant women: Not MPXV infected pregnant women
  Interventions: Other: routine care

INTERVENTIONS:
Other: routine care — routine care

SUMMARY:
PREGMPOXCO study addresses the escalating Mpox virus (MPXV) infections among pregnant women in South Kivu, DRC following a novel MPXV sub-lineage, predominantly transmitted through heterosexual contact, stressing critical gaps in our understanding of MPXV's impact on pregnant populations. To better understand this altered transmission pattern of MPXV and its impact on this vulnerable population, PREGMPOX will employ both passive and active surveillance techniques to methodologically capture MPXV incidence among pregnant women over two years, integrating data from routine antenatal care and targeted community outreach to timely assess the MPXV's effects on maternal and neonatal health. In sentinel study sites in hot spot areas, the incidence of mpox among pregnant women will be investigated and potential transmission routes determined. MPXV(+) pregnant women will be asked to participate in a cohort study where they will be followed until delivery to document pregnancy outcomes (e.g.: miscarriage, stillbirths, preterm deliveries, neonatal mpox), maternal immune response, virus abundance and pathological changes in the placenta. This will help to determine specific risk factors and modes and frequencies of vertical transmission to the unborn, and generate a list of clinical and immunological predictors for adverse outcomes for pregnant women and neonates. Data on MVA-BN exposure will also be captured to report on its real world effectiveness. As a prerequisite to evaluate the safety of the MVA-BN vaccine and tecovirimat treatment in pregnant women according to the new DRC guidelines, we will establish a comprehensive register of adverse pregnancy outcomes, using a pharmacovigilance model to monitor and analyse adverse events following immunization and treatment. The results of our multidisciplinary studies will be crucial for developing guidelines and recommendations to manage mpox more effectively during pregnancy, and for potentially influencing global health policies.

DETAILED DESCRIPTION:
The PREGMPOX study employs a prospective cohort design enriched with a nested case-control component, adeptly tracking the dynamics of MPXV infection among pregnant women.

This approach incorporates a rigorous baseline data collection phase that enhances the understanding of initial disease presentation and risk factors associated with confirmed MPXV infection. Such detailed profiling at baseline is critical for identifying early disease characteristics and potential co-factors affecting outcomes. Further, follow-up and endline assessments are strategically planned to estimate the incidence of new infections and assess mother-child health outcomes in various groups: those testing positive versus negative for MPXV, vaccinated versus unvaccinated individuals, and comparisons between those treated with tecovirimat versus those who are not. This structured analysis allows for an in-depth evaluation of intervention effectiveness and safety. The study design also includes a test-negative case-control approach as a secondary analytical method. While not the primary focus-given the high specificity of PCR in confirming MPXV in over 90% of cases-this approach is valuable for confirming intervention effectiveness under natural conditions. This methodology is designed to avoid the ethical concerns often associated with randomized control trials in vulnerable populations, ensuring the feasibility and relevance of the study's outcomes. PREGMPOX employs a strategic combination of passive and active surveillance methods to comprehensively track the spread of MPXV among pregnant women, aiming to capture the full spectrum of the virus's impact. Passive surveillance is embedded into routine antenatal care, where healthcare providers systematically monitor and document MPXV symptoms, leveraging the existing healthcare infrastructure. This allows for the continuous collection of data within a clinical setting. In contrast, active surveillance extends beyond the confines of healthcare facilities, involving community health workers who engage directly with the community to identify and document MPXV cases that might not otherwise come to clinical attention. This includes setting up specialized screening stations that facilitate the detection of cases in non-clinical environments. This dual surveillance approach is vital due to the severe risks associated with MPXV, particularly the high rates of foetal demise linked to severe infections. By combining both surveillance strategies, PREGMPOX enhances its capability for early detection and effective response, including prompt referral for necessary interventions. This comprehensive data collection and proactive case finding strategy are crucial for implementing timely interventions that could prevent severe outcomes in pregnant women and their foetuses, thereby mitigating the broader impact of the MPXV outbreak. PREGMPOX will also contribute to basic research in this vulnerable population where data is scarce by conducting immunological and histopathological assessments to understand the mechanisms underlying the impact of MPVX infection on pregnancy. These assessments will be conducted through a nested case-control study within the larger cohort. Samples will be collected at specific time points to evaluate immune responses to MPVX infection or vaccination and to study placental pathology in infected cases.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnancy status: all women confirmed to be pregnant at the time of recruitment.

  2. Age: women of all age (ascent to be asked for non-legal age to allow for the pair mother-child to benefit with earlier diagnosis and other befit the study might offer).

  3. Geographical inclusion: residing within the catchment areas of the selected healthcare facilities in South Kivu to ensure that they are likely to continue receiving follow-up care at the participating sites throughout their pregnancy.

  4. Symptomatic and asymptomatic participation:
  * Symptomatic: pregnant women presenting with symptoms suggestive of mpox, such as fever, rash/skin lesion, or lymphadenopathy.
  * Asymptomatic: pregnant women attending routine antenatal visits who do not exhibit symptoms but are screened as part of the study's surveillance efforts or who report a confirmed case of mpox in the household/or among closed contacts 5. Consent: women who provide written informed consent to participate in the study, having understood the purpose, procedures, potential risks, and benefits of the study.

Exclusion Criteria:1. Non-consent: pregnant women who do not consent/or their parent-caregiver to participate in the study.

2. Medical exclusions: women with pre-existing medical conditions that, as determined by clinical judgment, may either put them at risk due to participation in the study or could confound the study results (e.g., conditions that significantly alter immune response such as confirmed cancer).

3. Plans to relocate: women who plan to move out of the geographical study area during the study period, which would interfere with follow-up.

4. Participation in other studies: women currently participating in other clinical trials that might interfere with the results of this study, especially trials involving new experimental treatments for mpox or other infectious diseases.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women in the South Kivu province of the DRC at risk for mpox
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy outcome | at delivery
  health of the mother and child

IPD SHARING:
Plan to Share IPD: Undecided